CLINICAL TRIAL: NCT06122155
Title: Investigating How Cortical Modulation of the Cerebellum and Posterior Parietal Cortex Using Anodal tDCS Influences Ankle Motor Adaptation After Motor Learning
Brief Title: Effects of Posterior Parietal Cortex and Cerebellum Anodal tDCS on Ankle Tracking Visuomotor Adaptation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 202204075DINB
Record Dates: First submitted 2023-10-29; First posted 2023-11-08 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2022-05

CONDITIONS: Transcranial Direct Current Stimulation
Keywords: Transcranial Direct Current Stimulation
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Posterior parietal cortex (PPC) (Experimental): In the motor adaptation phase, a 20-minute, 2 mA anodal tDCS was delivered through two 5cm x 7cm electrodes using the DC-STIMULATOR MR (neuroConn, Germany). The electrical current gradually ramps up and down in 20 seconds. In the PPC group, the anodal electrode was placed over the P3 or P4 areas on the skull, covering the PPC area on the opposite side of the testing foot (according to the international 10-20 EEG system), and the reference electrode was placed over the supraorbital region on the same side of the testing foot.
  Interventions: Device: Transcranial direct current stimulation (Anodal)
- Cerebellum (Experimental): In the motor adaptation phase, a 20-minute, 2 mA anodal tDCS was delivered through two 5cm x 7cm electrodes using the DC-STIMULATOR MR (neuroConn, Germany). The electrical current gradually ramps up and down in 20 seconds. In the cerebellum group, the anodal electrode was placed 1~2 cm under and 3~4 cm lateral to the inion on the same side of the testing foot, with the reference electrode placed on the buccinator on the same side of the testing foot.
  Interventions: Device: Transcranial direct current stimulation (Anodal)
- Sham (Sham Comparator): In the motor adaptation phase, a 20-minute, 0 mA anodal tDCS was delivered through two 5cm x 7cm electrodes using the DC-STIMULATOR MR (neuroConn, Germany) for the sham group. Participants were informed that they might experience itchiness, burning, or mild discomfort during the tDCS period regardless of which group they were assigned to, so they would not use their sensation as a basis for determining whether they received actual stimulation or not.
  Interventions: Device: Transcranial direct current stimulation (Sham)

INTERVENTIONS:
Device: Transcranial direct current stimulation (Anodal) — 20-minutes, 2 mA anodal tDCS delivering through two 5 cm x 7 cm electrodes
  Arms: Cerebellum; Posterior parietal cortex (PPC)
Device: Transcranial direct current stimulation (Sham) — 20-minutes, 0 mA anodal tDCS delivering through two 5 cm x 7 cm electrodes
  Arms: Sham

SUMMARY:
Motor adaptation is guided by state estimation, a dynamic prediction of the interaction consequences between body and environment in the sensorimotor system. Previous studies have shown that the posterior parietal cortex (PPC) and cerebellum are potential candidates for state estimators. However, neither direct evidence linking neural substrates of state estimation and motor adaptation nor the differences in state estimation in these two brain areas was presented. A comparison of neuromodulation effects over PPC and cerebellum in motor adaptation tasks could provide direct evidence to solve the knowledge gap.

Objective: This study aims to provide direct evidence to link state estimation and motor adaptation, and the neuromodulation effects of PPC and cerebellum in motor adaptation by using anodal transcranial direct current stimulation.

DETAILED DESCRIPTION:
This was a single-blind, sham-controlled study. All participants were randomized to the PPC, cerebellum, and sham stimulation group. The ankle tracking system was used to record the ankle tracking visuomotor task during the motor learning phase, motor adaptation phase, and motor re-adaptation phase. Normalized root-mean squared error (RMSE) and RMSE reduction rate were measured as the performance outcome. A 20-minute atDCS at 2 mA anodal tDCS was given during the motor adaptation phase. The immediate effect and after effect of tDCS were seen in the motor adaptation phase and motor re-adaptation phase, respectively.

ELIGIBILITY:
Inclusion Criteria:

* age between 20~29 years old
* normal ankle range of motion and muscle strength
* intact cognitive function (Mini-mental State Examination (MMSE) >27)
* corrected vision > 0.9.

Exclusion Criteria:

* any neurologic or psychiatric disease history
* musculoskeletal disease that interferes lower extremities movement
* severe cardiopulmonary or systematic disease (e.g. unstable angina, severe arrhythmia, heart failure, hypertrophic cardiomyopathy, aortic stenosis, pulmonary embolism, kidney failure)
* paresthesia
* seizure history
* brain surgery, meningitis, encephalitis history
* drainage tube on the head
* metal or other insertion in the brain
* insertion of electric medical device (e.g. pacemaker, cochlear implant)
* pregnancy
* taking central nervous system medication (e.g. antidepressants, anxiolytic)
* alcoholic addiction or drug abuse
* open wound, allergy, rash, or other illness that would affect the placement of tDCS
* headache, disgusting, vomit, or any other severe side effect to the tDCS

Ages: 20 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-11-26 (Actual); Primary Completion 2023-06-19 (Actual); Study Completion 2023-06-19 (Actual)

PRIMARY OUTCOMES:
Block root-mean squared error (RMSE) | 2 hours during the time of assessment of the participant
  RMSE is the error between target trajectory and subject cursor trajectory. Every 5 trials of RMSE were averaged into one block.
RMSE reduction rate | 2 hours during the time of assessment of the participant
  ΔRMSEi-(i+1) = (RMSEi - RMSEi+1) / RMSEi x 100%

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
undecided